CLINICAL TRIAL: NCT00774683
Title: A Phase IV, Open-Label, Single-Sequence Pilot Study to Characterize the Pharmacokinetics of a 400mg Oral Dose of Raltegravir in the Cervicovaginal Fluids of HIV-Infected Women
Brief Title: A Pilot Study to Characterize the Pharmacokinetics of Raltegravir in the Cervicovaginal Fluids of HIV-infected Women
Status: Completed | Type: Observational
Sponsor: Kristine Patterson, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Kristine Patterson, MD, Clinical Associate Professor, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Other Study IDs: CID 0706 Sub-study A
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: HIV; AIDS
Keywords: Pilot; Pharmacokinetics; Raltegravir; Cervicovaginal; HIV; Women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood specimens and cervicovaginal fluids
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sub-study Group A: Six HIV-positive African American women from the main study, CID 0706
  Interventions: Drug: Raltegravir (Isentress®)

INTERVENTIONS:
Drug: Raltegravir (Isentress®) — 400 mg p.o. BID x 7 days
  Other Names: ISENTRESS; MK-0518

SUMMARY:
The purpose of this research sub-study is to learn about the levels of an antiretroviral (ARV) medication called Raltegravir, and response to HIV virus in the genital tract of HIV-positive women.

We would like to see how this study medication is tolerated, and how the body processes the study medication in women who are HIV-positive. More specifically, we are interested in how Isentress® might penetrate into the female cervicovaginal secretions thereby potentially reducing the amount of HIV in those secretions. A reduction in the amount of HIV in genital secretions may prevent female subjects from transmitting HIV to their sexual partners. This information will help the research team know how a medication such as Isentress® might be used to prevent the sexual transmission of HIV.

DETAILED DESCRIPTION:
Purpose: This study aims to characterize the pharmacokinetics of raltegravir in cervicovaginal fluids of HIV-infected women, and compare this to the blood plasma pharmacokinetics being obtained in the main study, CID 0706.

Participants: Six HIV-positive women from the CID 0706 study Procedures: During the pharmacokinetic visit to obtain blood plasma in the CID 0706 study, women will be asked to self-collect cervicovaginal samples using a vaginal aspirator at the following timepoints: pre-dose and 1, 2, 4, 6, 8, and 12 hours after raltegravir 400mg dose administration.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection documented by HIV serology or detectable viral load
* Self-described as African-American
* Less than 7 days cumulative of prior HIV therapy
* Plasma HIV RNA PCR equal to or greater than 1000 copies/mL within 90 days prior to study entry
* Able to provide informed consent
* In the opinion of the investigator, able to comply with study medication and procedures
* ALT (SGPT) < or equal to 3.0 x ULN within 45 days prior to study entry
* GRF > 60 as calculated by MDRD within 45 days prior to study entry
* All women of reproductive potential (who have not reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation) must have a negative serum or urine β-HCG pregnancy test performed within 48 hours before entry.

All study volunteers must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) and, if participating in sexual activity that could lead to pregnancy, the female study volunteer/male partner must use at least one reliable method of contraception (e.g., condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an IUD; or hormonal-based contraception), simultaneously while receiving the protocol-specified medication(s) and for 6 weeks after stopping the medication(s).

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Prior receipt of Raltegravir
* Any condition which in the opinion of the investigator is likely to interfere with follow-up or ability to take the study medication appropriately
* A positive test for bacterial vaginosis, syphilis, gonorrhea, Chlamydia, HSV-2 (active lesions), or trichomonas at entry or week 2 of the main study, CID 0706

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: UNC ID Clinic, Durham County Health Department, Wake County Health Department
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of raltegravir in cervicovaginal fluids of HIV-infected women, and compare this to the blood plasma pharmacokinetics being obtained in the main study, CID 0706. | Single Time Point Measurement at 4 Weeks after ART Initiation

CONTACTS AND LOCATIONS:
Overall Officials: Kristine B Patterson, MD, Principal Investigator — University of North Carolina, Chapel Hill; Angela DM Kashuba, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Musicco M, Lazzarin A, Nicolosi A, Gasparini M, Costigliola P, Arici C, Saracco A. Antiretroviral treatment of men infected with human immunodeficiency virus type 1 reduces the incidence of heterosexual transmission. Italian Study Group on HIV Heterosexual Transmission. Arch Intern Med. 1994 Sep 12;154(17):1971-6. PMID 8074601
- [Background] Otten RA, Smith DK, Adams DR, Pullium JK, Jackson E, Kim CN, Jaffe H, Janssen R, Butera S, Folks TM. Efficacy of postexposure prophylaxis after intravaginal exposure of pig-tailed macaques to a human-derived retrovirus (human immunodeficiency virus type 2). J Virol. 2000 Oct;74(20):9771-5. doi: 10.1128/jvi.74.20.9771-9775.2000. PMID 11000253
- [Background] Lallemant M, Jourdain G, Le Coeur S, Mary JY, Ngo-Giang-Huong N, Koetsawang S, Kanshana S, McIntosh K, Thaineua V; Perinatal HIV Prevention Trial (Thailand) Investigators. Single-dose perinatal nevirapine plus standard zidovudine to prevent mother-to-child transmission of HIV-1 in Thailand. N Engl J Med. 2004 Jul 15;351(3):217-28. doi: 10.1056/NEJMoa033500. Epub 2004 Jul 9. PMID 15247338
- [Background] Blankson JN, Persaud D, Siliciano RF. The challenge of viral reservoirs in HIV-1 infection. Annu Rev Med. 2002;53:557-93. doi: 10.1146/annurev.med.53.082901.104024. PMID 11818490
- [Background] Pierson T, Hoffman TL, Blankson J, Finzi D, Chadwick K, Margolick JB, Buck C, Siliciano JD, Doms RW, Siliciano RF. Characterization of chemokine receptor utilization of viruses in the latent reservoir for human immunodeficiency virus type 1. J Virol. 2000 Sep;74(17):7824-33. doi: 10.1128/jvi.74.17.7824-7833.2000. PMID 10933689
- [Background] Markowitz M, Morales-Ramirez JO, Nguyen BY, Kovacs CM, Steigbigel RT, Cooper DA, Liporace R, Schwartz R, Isaacs R, Gilde LR, Wenning L, Zhao J, Teppler H. Antiretroviral activity, pharmacokinetics, and tolerability of MK-0518, a novel inhibitor of HIV-1 integrase, dosed as monotherapy for 10 days in treatment-naive HIV-1-infected individuals. J Acquir Immune Defic Syndr. 2006 Dec 15;43(5):509-15. doi: 10.1097/QAI.0b013e31802b4956. PMID 17133211
- [Background] Cohen MS. Preventing sexual transmission of HIV. Clin Infect Dis. 2007 Dec 15;45 Suppl 4:S287-92. doi: 10.1086/522552. PMID 18190301
- [Background] Isentress (Raltegravir) Prescribing Guide. Merck & Co., Inc. October 2007